CLINICAL TRIAL: NCT02762448
Title: Interferon-free Antiviral Treatment of HCV-Positive Genotype 1b Related Indolent Non-Hodgkin Lymphomas Patients Using Daclatasvir and Asunaprevir: A Pilot Study
Brief Title: Interferon-free Antiviral Treatment of HCV-Positive Genotype 1b Related Indolent Non-Hodgkin Lymphomas
Status: Withdrawn | Type: Observational
Why Stopped: no patient enrollment
Sponsor: Tainan Municipal Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AI447-122
Record Dates: First submitted 2016-04-28; First posted 2016-05-05 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis c
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Daclatasvir + Asunaprevir: Prospectively collect cases with NHL (n=10), having HCV genotype 1b related NHL, who will be treated with ASV (200 mg twice daily) + DCV(60 mg once daily) for 24 weeks .
  Interventions: Drug: Daclatasvir+ Asunaprevir

INTERVENTIONS:
Drug: Daclatasvir+ Asunaprevir — HCV clearance and complete regression of NHL by ASV+ DCV
  Other Names: DCV;ASV

SUMMARY:
Interferon-free Antiviral Treatment of HCV-Positive Genotype 1b Related Indolent non-Hodgkin Lymphomas Patients Using Daclatasvir and Asunaprevir: A Pilot Study

DETAILED DESCRIPTION:
Prospectively collect cases with NHL (n=10), having HCV genotype 1b related NHL, who will be treated with ASV (200 mg twice daily) + DCV(60 mg once daily) for 24 weeks The patients will be observed and followed to determine whether there is regression of NHL after antiviral treatment. Conventional chemotherapy should be initiated shortly in cases without regression.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. 18 to 70 years of age
3. Who had chronic HCV genotype 1b infection
4. An HCV RNA level of 105 IU per milliliter or higher
5. Being diagnosed to be low grade B cell non-Hodgkin lymphoma

Exclusion Criteria:

1. Patients with hepatitis B virus infection,
2. Other liver diseases
3. HIV infection,
4. Pre-existing HCV variants in the NS5A domain included Q30R, L31 M/V, and Y93C/N
5. Evidence of cirrhosis, as documented by means of either liver biopsy or assessment of imaging results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an open label pilot without control group or other intervention. Participants will be recruited to a known intervention. Assessments will be conducted in an unblinded fashion. In terms of genotypes, 1b and 2a were suggested to be risk factors for the developing lymphoma in most HCV patients. In HCV-infected patients with splenic marginal zone or indolent B-cell NHL, many studies reported that combined treatment with interferon-alpha and ribavirin may lead to HCV clearance and concomitant regression of lymphomas
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
HCV clearance and complete regression of NHL by ASV+ DCV | 2years
  patients who had undetectable HCV RNA levels at or after week 4. Viral relapse was defined as confirmed detectable HCV RNA levels during the post-treatment follow-up period in patients who had had undetectable HCV RNA levels at the end of treatment

IPD SHARING:
Plan to Share IPD: Undecided